CLINICAL TRIAL: NCT06191939
Title: Adapting and Testing a Novel Self-Compassion Intervention to Reduce Lung Cancer Stigma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola Marymount University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Timothy Williamson, Assistant Professor, Loyola Marymount University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LMU IRB 2022 SU 27-R; R00CA256351 (NIH)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: stigma; self-compassion; pilot; adaptation
MeSH Terms: conditions — Lung Neoplasms; Social Stigma | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindful Self-Compassion for Lung Cancer (MSC-LC) (Experimental): Group-based psychosocial intervention adapted from Mindful Self-Compassion that focuses on the development of mindfulness and self-compassion skills to reduce lung cancer stigma.
  Interventions: Behavioral: Mindful Self-Compassion for Lung Cancer (MSC-LC)
- Enhanced standard of care with waitlist (Active Comparator): Control group that will receive a list of mental health resources and will complete questionnaire assessments during a parallel timeframe as participants in the intervention condition and be placed on a waiting list to receive the MSC-LC intervention after study completion.
  Interventions: Other: Enhanced standard of care with waitlist

INTERVENTIONS:
Behavioral: Mindful Self-Compassion for Lung Cancer (MSC-LC) — The overall goal of this 10-week, group-based, virtually-delivered, psychosocial intervention is to enhance recognition and responsiveness to difficult thoughts and emotions and to build self-compassion skills that facilitate patients' ability to turn inward to those thoughts and feelings with mindfulness, connectedness, and self-kindness. Each weekly session is designed to be 90 minutes and follows an agenda with highly structured scripts covering self-compassion topics (e.g., pain of disconnection, listening with compassion), which are carefully organized to build upon one another. In each session, didactic topics (e.g., "What is self-compassion?") taught by trained interventionists lead into guided experiential learning practices (e.g., guided meditation), which are then followed by inquiry into the participants' direct experiences of the practices. The treatment manual is adapted based on the Mindful Self-Compassion Teacher Guide (from the Center for Mindful Self-Compassion).
  Arms: Mindful Self-Compassion for Lung Cancer (MSC-LC)
Other: Enhanced standard of care with waitlist — Participants in the enhanced standard of care control condition will be provided with an information sheet from the NCI about how to find helpful organizations and resources in their community. Self-report will be used to describe any supportive care services pursued by the participant. Additionally, control participants will be added to a waiting list for receiving the MSC-LC intervention program. After completing all questionnaire assessments (16 weeks following study entry), the study team will offer the MSC-LC intervention program to participants on the waiting list.
  Arms: Enhanced standard of care with waitlist

SUMMARY:
The goal of this pilot clinical trial is to test a disease-tailored, mindfulness-based intervention (Mindful Self-Compassion for Lung Cancer; MSC-LC) in adults diagnosed with lung cancer who are experiencing stigma. The current project seeks to:

* Evaluate preliminary evidence for the feasibility, acceptability, and preliminary efficacy of MSC-LC in reducing stigma for adults with lung cancer, compared to a waitlist control condition
* Elicit interventional impact not captured through quantitative measures with qualitative data from purposively sampled high responders and non-responders from the intervention condition

Participants will randomized to either the MSC-LC intervention (a 10-week, virtually-delivered, group-based psychosocial intervention focused on the development of mindfulness and self-compassion skills) or to a waitlist control group that receives a referral to an NCI list of helpful mental health resources in their community. Researchers will compare the intervention and control groups to see if the MSC-LC intervention reduces lung cancer stigma and increases self-compassion.

DETAILED DESCRIPTION:
Lung cancer stigma (i.e., perceived and internalized negative appraisal and devaluation associated with lung cancer) is a pervasive problem experienced by the majority of lung cancer patients. Notably, experiences of lung cancer stigma are strongly associated with poorer quality of life and higher depressive symptoms. Despite these associations, there is a gap in the field regarding empirically supported, patient-focused interventions that target the reduction of lung cancer stigma.

Self-compassion (i.e., directed kindness towards oneself in times of suffering) is a protective psychosocial factor that has been targeted through intervention approaches to reduce shame and self-criticism in non-cancer samples. Additionally, higher self-compassion has been shown to attenuate the relationship between lung cancer stigma and depression, suggesting that fostering self-compassion may be an effective intervention strategy to reduce lung cancer stigma. Mindful Self-Compassion is an empirically supported, 8-week psychosocial intervention demonstrated to increase self-compassion and reduce feelings of shame, distress, depression, and anxiety in non-cancer samples. However, given several anticipated challenges associated with delivering Mindful Self-Compassion to lung cancer patients (e.g., breathing challenges that arise during breath-focused meditations, fatigue that interferes with attending 3-hour sessions), the investigators developed an adapted version of the intervention (Mindful Self-Compassion for Lung Cancer; MSC-LC) that is tailored to the needs of adults diagnosed with lung cancer, addresses delivery challenges, and targets the reduction of lung cancer stigma.

This is a pilot trial examining the feasibility, acceptability, and preliminary efficacy of MSC-LC, compared to waitlist control condition. The central hypothesis is that MSC-LC will be demonstrate high feasibility and acceptability as well as preliminary efficacy in reducing lung cancer stigma and promoting self-compassion.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age as per self report;
* Has a confirmed lung cancer diagnosis, as per self-report and confirmed by clinician judgment or medical record note;
* Endorses elevated levels of lung cancer stigma (scores >37.5 on the Lung Cancer Stigma Inventory)
* Able to read and respond to questions in English

Exclusion Criteria:

* Inability to understand study procedures or informed consent process, or significant personality dysfunction likely to interfere with study participation, as per study clinician's judgment
* Completed a course of Mindful Self-Compassion or an equivalent meditation training in the last year
* Use of antidepressant, anxiolytic, antipsychotic, or mood stabilizing medication(s) for which the dose has been initiated or changed within the 8 weeks prior to study entry

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer Stigma Inventory | Study Entry, 5 weeks (mid-intervention), 10 weeks (post-intervention; primary outcome), 16 weeks (long-term follow-up)
  The Lung Cancer Stigma Inventory is a self-report questionnaire of lung cancer stigma, which includes 25 items rated on a 5-point Likert scale. Scores range from 25-125, with higher scores indicating higher lung cancer stigma.

SECONDARY OUTCOMES:
Patient Health Questionnaire-8 | Study Entry, 5 weeks (mid-intervention), 10 weeks (post-intervention), 16 weeks (long-term follow-up)
  The Patient Health Questionnaire-8 is a self-report questionnaire of depressive symptoms, which includes 8 items rated on a 4-point Likert scale. Scores range from 0-24, with higher scores indicating higher depressive symptoms.
Generalized Anxiety Disorder-7 | Study Entry, 5 weeks (mid-intervention), 10 weeks (post-intervention), 16 weeks (long-term follow-up)
  The Generalized Anxiety Disorder-7 is a self-report questionnaire of anxiety symptoms, which includes 7 items rated on a 4-point Likert scale. Scores range from 0-21, with higher scores indicating higher anxiety symptoms.
Self-Compassion Scale | Study Entry, 5 weeks (mid-intervention), 10 weeks (post-intervention), 16 weeks (long-term follow-up)
  The Self-Compassion Scale is a self-report questionnaire of self-compassion, which includes 26 items rated on a 5-point Likert scale. Scores range from 26-130, with higher scores indicating higher self-compassion.
Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being, meaning and peace subscales | Study Entry, 5 weeks (mid-intervention), 10 weeks (post-intervention), 16 weeks (long-term follow-up)
  The Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being is a self-report questionnaire on meaning and peace, which includes 8 items rated on a 5-point Likert scale. Scores range from 0-48, with higher scores indicating higher self-reported meaning and peace during chronic illness.

OTHER OUTCOMES:
Number of intervention sessions that each consented participant attended | 10 weeks (post-intervention)
  This measure will be calculated as a count of sessions that each consented participant in the MSC-LC intervention attended. It will be used as a metric of acceptability of the intervention.
Treatment fidelity | Weekly throughout the intervention from study entry to post-intervention (10 weeks)
  This measure will be calculated as a proportion of the number of components within an intervention session that the interventionists delivered (assessed via audio recording) over the number of pre-determined components that they were meant to deliver, per the interventionist manual.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Williamson, Ph.D., MPH, Principal Investigator — Loyola Marymount University
Locations (1):
- Loyola Marymount University, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Loyola Marymount University supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication.
Access Criteria: Requests may be made to: timothy.williamson@lmu.edu